CLINICAL TRIAL: NCT02296086
Title: A Prospective Multicenter Cohort Study to Evaluate the Effect of Early Mobilization of Patients After Hip Fracture Fixation on Functional Outcomes in the Chinese Population
Brief Title: MobiChina - A Prospective Multicenter Cohort Study
Status: Completed | Type: Observational
Sponsor: AO Innovation Translation Center (Other)
Responsible Party: Sponsor
Other Study IDs: MobiChina
Record Dates: First submitted 2014-11-14; First posted 2014-11-20 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2019-09

CONDITIONS: Unstable Fracture; Hip Fracture
Keywords: Geriatrics [MeSH]; Hip fractures [MeSH]; China [MeSH]; Early ambulation [MeSH]; Immobilization [MeSH]
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group I: Study sites in which patients perform early mobilization as per local standard of care, which is as follows:
  * 2 days (at the latest) after surgery: Transfer from the bed to a sitting chair for the first time
  * 4 (± 2) days after surgery: Stand up and put both feet on the ground for the first time (walking aids allowed)
  * 5 (± 2) days after surgery: Walking (at least partial weight bearing, walking aids allowed)
  * The patients are instructed by the investigator at the hospital about a standardized mobilization program to be followed at home
- Group II: Study sites in which patients start walking (i.e. partial weight bearing, walking aids allowed) more than 7 days after surgery as per local standard of care

SUMMARY:
The study will assess the difference in functionality between early vs. standard mobilization after hip fracture in the Chinese population.

DETAILED DESCRIPTION:
The primary objective of this prospective observational cohort study is to assess the difference in functionality between Group I and II (see mobilization regimens for the two groups above) at 6 weeks using the modified Barthel Index in the Chinese population.

The allocation of patients to the two groups will be performed on a clinic level: 50% of patients will be recruited by study sites in Group I (early mobilization). The other 50% of patients will be recruited by study sites in Group II. The sites are carefully selected after evaluating their standard procedures of mobilizing elderly patients after hip fractures. This process is documented using formal site selection questionnaires.

The modified Barthel Index is estimated at 75 points for Group II and at 85 points for Group I.

Patients aged 65 years and older with unstable intertrochanteric fractures (AO 31 A2 or A3) treated with an intramedullary nail will be included in this study.

The study visits will be defined as preoperative, surgery, discharge, 6 (± 2) weeks and 12 (± 2) weeks follow-up (FU) visits. Furthermore, there will be a telephone contact 12 months (± 1 month) postsurgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 and older
* Diagnosis of an unstable intertrochanteric fractures (AO 31- A2 or A3) treated with an intramedullary nail
* Ability to walk independently or with a walking aid prior to injury
* Informed consent obtained, i.e.: Ability of the patient to understand the content of the patient information / Informed Consent Form and signed and dated Institutional Review Board (IRB) / Ethics Committee (EC)-approved written informed consent

Exclusion Criteria:

* Severe dementia
* Recent history of substance abuse (ie, recreational drugs, alcohol) that would preclude reliable assessment
* Prisoner
* Participation in any other medical device or medicinal product study within the previous month that could influence the results of the present study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 284 (Actual)
Dates: Start 2015-04; Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Modified Barthel Index | 6 weeks postoperative
  Investigator completed score

SECONDARY OUTCOMES:
Modified Barthel Index | Baseline
  Modified Barthel Index is retrospectively assessed for the pre-injury status using an investigator completed score
Modified Barthel Index | 12 weeks postoperative
  Investigator completed score
Immobilization-related adverse events | From surgery to 1 year follow-up
  Immobilization-related adverse events:
  * Pneumonia
  * Lung embolism
  * Pressure sores/ulcers
  * Urinary tract infections
Fixation failures | From surgery up to 1 year follow-up
  As assessed by the local investigator
Any other adverse events | From surgery up to 1 year follow-up
Mortality | From surgery up to 1 year postoperative
Muscle loss | From surgery up to 1 year follow-up
  Calf circumference measurement comparison: Loss calculated in %
Time to achieve partial and full weight bearing | From surgery to 1 year follow-up
  Will be assessed during the patient interview
Duration of hospital stay | For the duration of hospital stay, an expected average of 3 weeks
Numbers of re-admissions to the hospital | From surgery to 1 year follow-up
Quality of life: EuroQoL (EQ-5D) | 12 weeks postoperative
  Quality of life questionnaire using the EQ-5D
Residential status | Baseline to 1 year follow-up
  Will be assessed during the patient interview

CONTACTS AND LOCATIONS:
Overall Officials: Frankie Leung, MD, Principal Investigator — Queen Mary Hospital, Hong Kong
Locations (11):
- China (9):
  - JiShuiTan Hopsital, Beijing, Beijing Municipality
  - 3th Hospital of Hebei Medical University of Hebei, Hebei, Hebei
  - DCN Hospital, Beijing
  - West China Hospital of Sichuan University, Chengdu
  - Yunnan Second People Hospital, Kunming
  - Nantong University 1st Affiliated Hospital, Nantong
  - Shanghai Sixth People Hospital, Shanghai
  - The University of Hong Kong-Shenzhen Hospital, Shenzhen
  - Hong Hui Hospital, Xi'an
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong, Pokfulam
  - Queen Elisabeth Hospital, Hong Kong